CLINICAL TRIAL: NCT02503917
Title: Gynaecologic Organ Segmentation and Motion Tracking Using Ultrasound
Acronym: GENIUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4342
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Cervical Cancer
Keywords: Imaging, Ultrasound; Image-guided radiotherapy; Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy female adult volunteers
- Cervical cancer patients: Patients receiving radiotherapy for cervical cancer at the Royal Marsden who will receive a planning CT scan and daily CBCT scanning as part of their treatment.

SUMMARY:
This study will establish the feasibility and accuracy of localising and outlining the uterus on ultrasound images using both healthy volunteer and cervical patient cohorts. This will enable us to determine whether or not ultrasound will be a good option to ensure the correct patient position prior to radiotherapy for cervical cancer patients.

DETAILED DESCRIPTION:
Radiotherapy is an established and effective method for treating cancer, but it can have negative side effects if healthy tissues are also exposed to radiation. In the case of cervical cancer, the bladder, small bowel, and bone marrow are often irradiated, which can result in both short-term and long-term side effects. There are sophisticated radiation delivery techniques (known as IMRT and VMAT) which are capable of administering the radiation dose in a precise and controlled manner so that the intended target is irradiated and the healthy tissue is spared. However, the only way for these sophisticated radiation delivery methods to work in cervical cancer is to localise the uterus prior to radiotherapy treatment so that the lineup between the radiation beam and the target is ensured. The uterus is a relatively mobile organ, and can have very different positions within the body depending on the patient position, bladder volume, tumour site, etc. Currently, we are unable to take advantage of the sophisticated radiation delivery techniques as we have no reliable way of seeing where the uterus is. Ultrasound is a promising way to overcome this problem.

Ultrasound is non-ionising, has good soft-tissue contrast, and can easily be incorporated into the radiation treatment room. We wish to establish the feasibility and accuracy of localising and outlining the uterus on ultrasound images. This will enable us to determine whether or not ultrasound will be a good option to ensure the correct patient position prior to radiotherapy for cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer cohort: Healthy female adult volunteers
* patient volunteer cohort: Patients receiving radiotherapy for cervical cancer who will receive a planning CT scan and daily CBCT scanning as part of their treatment.

Exclusion Criteria:

* both cohorts: Women who have received hysterectomies and women who are pregnant at the time of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteer cohort: Healthy female adult volunteers patient volunteer cohort: Patients receiving radiotherapy for cervical cancer who will receive a planning CT scan and daily CBCT scanning as part of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of ultrasound scans with dice similarity coefficient (DSC) of >0.90 between algorithm-derived contour and ground-truth contour | DSC calculated at 24 time points for each healthy volunteer (3 days)
  The DSC between the ground truth contour and the algorithm derived contour will indicate the accuracy of the segmentation algorithm.
Coefficient of variation between of expert-drawn contours on ultrasound and expert-drawn contours on CBCT | COV calculated at a minimum of 3 time points during 6 weeks that the patient is receiving radiation therapy
  A small COV will indicate greater clinician/expert confidence in segmenting the uterus

SECONDARY OUTCOMES:
Bland-Altman plot (healthy volunteer cohort) | 1 day
  Used to describe the level of agreement between MR and ultrasound images of the uterus.
Uterine center of mass displacement on ultrasound (healthy volunteer cohort) | 3 days
  Assess both inter- and intra- fractional motion of the uterus.
Expert confidence scores for each imaging modality (ultrasound and MR) (healthy volunteer cohort) | from data collected over 3 days
  Determine if uterine segmentation on ultrasound receives acceptable confidence score compared with MR
Bland-Altman plot (patient volunteer cohort) | 6 weeks
  describe level of agreement among the COV, circularity index, volume, and centre of mass position betweeen ultrasound, CT, and CBCT.
Expert confidence scores for each imaging modality (ultrasound, CT, and CBCT) (patient volunteer cohort) | from data collected over 6 weeks
  Determine if uterine segmentation on ultrasound receives greater confidence score compared with CT and CBCT.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lalondrelle, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey, United Kingdom